CLINICAL TRIAL: NCT04301791
Title: the Impact of Nutritional Status on Clinical Outcome of Children Admitted in PICU OF Assuit Children University Hospital
Brief Title: Impact of Nutritional Status on Clinical Outcome in PICU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hager Adel Ali, principal investigator, Assiut University
Other Study IDs: nutritional status
Record Dates: First submitted 2020-03-01; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Nutritional Disorder
MeSH Terms: conditions — Nutrition Disorders | interventions — Nutritional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: nutritional status — impact of nutritional status on clinical outcome of children admitted in PICU

SUMMARY:
Malnutrition is believed to be associated with clinical outcomes in ill patients and several studies have shown that nutrition status play a major role in disease prognosis in adults .

Different authors have described an increase in morbidity and mortality attributable to malnutrition, as it lead to state of partial immunosuppression, delay wound healing ,causes muscular atrophy and increase length of stay.

DETAILED DESCRIPTION:
Several studies have investigated the predictive role of an extremely low body weight on disease prognosis and outcomes among general and critically ill children .They enrolled all patients consecutively admitted to pediatric intensive care unit PICU) , therefore , being underweight may have resulted from endocrine diseases, genetic syndromes or other systemic underlying illnesses .

The impact of low body weight on outcomes of acutely critically ill but previously healthy children is still unknown.

Many studies evaluate the clinical status and outcome by pediatric index of mortality (PIM2) as a popular and reliable predictive score .

In this study, we will investigate the impact of being underweight or proper weight on mortality and morbidity among acute critically ill children with no genetic, endocrine, or chronic systemic illness at PICU admission

ELIGIBILITY:
Inclusion Criteria:

1. All children admitted to PICU with nutritional disorders
2. Children with acute diseases and anthropometric measurements taken within first 24hours

Exclusion Criteria:

1-children with underlying chronic diseases (eg cerebral palsy ,type 1 or 2 diabetes , epilepsy, metabolic diseases, inflammatory bowel disease , liver cirrhosis , immunodeficiency , autoimmune disordes , malignancy , chronic kidney disease) and postoperative patients.

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: children age from one month to 18 years with no chronic diseases admitted at PICU at Assiut university hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
the correlation between nutritional status of children admitted in PICU and outcomes | 2 years
  nutritional status measured by weight in kilograms and height in meters will be combined to report BMI for Z scoreand outcomes measured by pediatric index of mortality2 (PIM2)

REFERENCES:
- [Background] Calle EE, Thun MJ, Petrelli JM, Rodriguez C, Heath CW Jr. Body-mass index and mortality in a prospective cohort of U.S. adults. N Engl J Med. 1999 Oct 7;341(15):1097-105. doi: 10.1056/NEJM199910073411501. PMID 10511607
- [Background] Marcos A, Nova E, Montero A. Changes in the immune system are conditioned by nutrition. Eur J Clin Nutr. 2003 Sep;57 Suppl 1:S66-9. doi: 10.1038/sj.ejcn.1601819. PMID 12947457
- [Background] Hulst J, Joosten K, Zimmermann L, Hop W, van Buuren S, Buller H, Tibboel D, van Goudoever J. Malnutrition in critically ill children: from admission to 6 months after discharge. Clin Nutr. 2004 Apr;23(2):223-32. doi: 10.1016/S0261-5614(03)00130-4. PMID 15030962
- [Background] Kielmann AA, McCord C. Weight-for-age as an index of risk of death in children. Lancet. 1978 Jun 10;1(8076):1247-50. doi: 10.1016/s0140-6736(78)92478-9. PMID 78007
- [Background] Numa A, McAweeney J, Williams G, Awad J, Ravindranathan H. Extremes of weight centile are associated with increased risk of mortality in pediatric intensive care. Crit Care. 2011;15(2):R106. doi: 10.1186/cc10127. Epub 2011 Mar 31. PMID 21453507
- [Background] Bagri NK, Jose B, Shah SK, Bhutia TD, Kabra SK, Lodha R. Impact of Malnutrition on the Outcome of Critically Ill Children. Indian J Pediatr. 2015 Jul;82(7):601-5. doi: 10.1007/s12098-015-1738-y. Epub 2015 Mar 26. PMID 25804317
- [Background] Czaja AS, Scanlon MC, Kuhn EM, Jeffries HE. Performance of the Pediatric Index of Mortality 2 for pediatric cardiac surgery patients. Pediatr Crit Care Med. 2011 Mar;12(2):184-9. doi: 10.1097/PCC.0b013e3181e89694. PMID 20581732
- [Background] Slater A, Shann F, Pearson G; Paediatric Index of Mortality (PIM) Study Group. PIM2: a revised version of the Paediatric Index of Mortality. Intensive Care Med. 2003 Feb;29(2):278-85. doi: 10.1007/s00134-002-1601-2. Epub 2003 Jan 23. PMID 12541154
- [Background] Prince NJ, Brown KL, Mebrahtu TF, Parslow RC, Peters MJ. Weight-for-age distribution and case-mix adjusted outcomes of 14,307 paediatric intensive care admissions. Intensive Care Med. 2014 Aug;40(8):1132-9. doi: 10.1007/s00134-014-3381-x. Epub 2014 Jul 18. PMID 25034475
- [Background] Mehta NM, Bechard LJ, Cahill N, Wang M, Day A, Duggan CP, Heyland DK. Nutritional practices and their relationship to clinical outcomes in critically ill children--an international multicenter cohort study*. Crit Care Med. 2012 Jul;40(7):2204-11. doi: 10.1097/CCM.0b013e31824e18a8. PMID 22564954
- [Background] Barker LA, Gout BS, Crowe TC. Hospital malnutrition: prevalence, identification and impact on patients and the healthcare system. Int J Environ Res Public Health. 2011 Feb;8(2):514-27. doi: 10.3390/ijerph8020514. Epub 2011 Feb 16. PMID 21556200
- [Background] Moreno Villares JM, Varea Calderon V, Bousono Garcia C, Lama More R, Redecillas Ferreiro S, Pena Quintana L; Sociedad Espanola de Gastroenterologia. [Nutrition status on pediatric admissions in Spanish hospitals; DHOSPE study]. Nutr Hosp. 2013 May-Jun;28(3):709-18. doi: 10.3305/nh.2013.28.3.6356. Spanish. PMID 23848094
- [Background] Cahill NE, Dhaliwal R, Day AG, Jiang X, Heyland DK. Nutrition therapy in the critical care setting: what is "best achievable" practice? An international multicenter observational study. Crit Care Med. 2010 Feb;38(2):395-401. doi: 10.1097/CCM.0b013e3181c0263d. PMID 19851094
- [Background] de Souza Menezes F, Leite HP, Koch Nogueira PC. Malnutrition as an independent predictor of clinical outcome in critically ill children. Nutrition. 2012 Mar;28(3):267-70. doi: 10.1016/j.nut.2011.05.015. Epub 2011 Aug 27. PMID 21872433
- See also: WHO Multicentre Growth Reference Study Group. WHO Child Growth Standards: Length/Height-for-Age, Weight-for-Age, Weight-for Length, Weight-for-Height and Body Mass Index-for-Age. Methods and Development. Geneva, Switzerland: World Health Organization — http://www.who.int/childgrowth/standards/technical_report/en/